CLINICAL TRIAL: NCT04537104
Title: Investigating Arrhythmias in a High-risk Population With Heart Failure Using Remote Monitoring (Coala Heart Monitor)
Brief Title: Remote Monitoring in Patients With Heart Failure
Acronym: REM-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Coala Life, Inc (Industry)
Responsible Party: Principal Investigator, Morten Lamberts, Associate Professor and Research Director, Herlev and Gentofte Hospital
Other Study IDs: P-2020-551
Record Dates: First submitted 2020-08-26; First posted 2020-09-03 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: arrhythmias; heart failure; remote monitoring
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Coala Heart Monitor — ECG monitoring

SUMMARY:
This study is a prospective cohort study with consecutive enrollment of newly diagnosed heart failure patients, investigating the prevalence and types of arrhythmias in this high-risk population using non-invasive remote monitoring with the Coala Heart Monitor. Participants are scheduled to use the Coala Heart Monitor twice daily or during symptoms (e.g. syncope, presyncope, palpitations, chest discomfort, or shortness of breath) to record a thumb and chest ECG over 3 months. Patient compliance with the recordings, self-reported health, response to technology, and experience using the device will additionally be assessed by self-developed questionnaires and the Kansas City Cardiomyopathy Questionnaire (KCCQ) at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Owns or has access to a smartphone
* Newly diagnosed moderate to severe heart failure (NYHA II-IV and left ventricular ejection fraction ≤ 40%)

Exclusion Criteria:

* Earlier atrial fibrillation/atrial flutter with indication for oral anticoagulant (OAC) treatment
* Pacemaker
* Cardiac resynchronization device
* Indications for OAC treatment (also low molecular weight heparin) due to atrial arrhythmias, mechanical heart valve, deep vein thrombosis, or pulmonary embolism.
* Expected survival ≤ 6 months
* Absolute contraindications for starting OAC treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed heart failure patients > 18 years of age from heart failure clinic
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
New-onset arrhythmias | 3 months
  Incidence of newly diagnosed atrial fibrillation/atrial arrhythmias on patient-activated thumb and chest ECG recordings

SECONDARY OUTCOMES:
Patient compliance | Week 8
  Patient compliance with at least two daily recordings.
Patient self-reported health | 3 months
  Patient self-reported health assessed by KCCQ.
Patient-reported outcomes | 3 months
  Patients' response to technology and experience using the device assessed by self-developed questionnaire.
Assessing recordings | 3 months
  Where there are interpretations of arrhythmias on recordings, agreement of recordings with subsequent Holter monitoring will be assessed.
Subsequent prescriptions | 3 years
  Through linkage with nationwide health care databases, subsequent prescription patterns of diuretics and antithrombotic medication in patients with and without atrial fibrillation.
Subsequent implantations | 3 years
  Through linkage with nationwide health care databases, subsequent implantation of cardiac devices in patients with and without atrial fibrillation.
Subsequent readmissions | 3 years
  Through linkage with nationwide health care databases, subsequent readmissions to hospital in patients with and without atrial fibrillation.
All-cause mortality | 3 years
  Through linkage with nationwide health care databases, all-cause mortality in patients with and without atrial fibrillation.
Cardiovascular mortality | 3 years
  Through linkage with nationwide health care databases, cardiovascular mortality in patients with and without atrial fibrillation.
Admissions for worsening heart failure | 3 years
  Through linkage with nationwide health care databases, and admission for worsening heart failure in patients with and without atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Herlev & Gentofte Hospital, Copenhagen, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided